CLINICAL TRIAL: NCT06519578
Title: Prospective Real-World Study of Hepatic Arterial Infusion Chemotherapy (HAIC) With Raltitrexed or 5-Fluorouracil for the Treatment of Hepatocellular Carcinoma
Brief Title: Prospective Real-World Study of HAIC With Raltitrexed or 5-Fluorouracil for the Treatment of Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Renji-LY2024-157-b
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX-HAIC Cohort (Other): Patients in this group received hepatic arterial infusion chemotherapy, with the following protocol:
  Oxaliplatin 85 mg/m^2
  Leucovorin calcium 400 mg/m^2
  Fluorouracil 400 mg/m^2 on Day 1, 2400 mg/m^2 continuous infusion for 46 hours
  Arterial infusion, once every 3 weeks
  Interventions: Drug: hepatic artery infusion chemotherapy
- RALOX-HAIC Cohort (Other): Patients in this group received hepatic arterial infusion chemotherapy, with the following protocol:
  Oxaliplatin 100 mg/m^2
  Raltitrexed 3 mg/m^2
  Arterial infusion, once every 3 weeks
  Interventions: Drug: hepatic artery infusion chemotherapy

INTERVENTIONS:
Drug: hepatic artery infusion chemotherapy — HAIC is a regional therapy that takes advantage of the fact that hepatic tumors, particularly hepatocellular carcinoma, predominantly receive their blood supply from the hepatic artery. The procedure typically involves the insertion of a catheter into the hepatic artery, often through a percutaneous approach or during a surgical procedure.
  FOLFOX (5-fluorouracil, leucovorin combined with oxaliplatin) or RALOX (raltitrexed combined with oxaliplatin) Q3W.
  Other Names: HAIC

SUMMARY:
This study is a prospective cohort study aimed at comparing the efficacy and safety of RALOX-HAIC and FOLFOX-HAIC in the treatment of hepatocellular carcinoma. It is planned to enroll 1115 patients with BCLC Stage B or C hepatocellular carcinoma, who will receive FOLFOX-HAIC or RALOX-HAIC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of clinically significant pleural effusion, ascites, or pericardial effusion that requires repeated treatment (puncture or drainage, etc.);
* History of immunodeficiency, including positive HIV test, or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Severe cardiovascular and cerebrovascular diseases, including but not limited to, myocardial infarction, severe/unstable angina, congestive heart failure (NYHA heart function classification ≥2), clinically significant supraventricular or ventricular arrhythmias requiring drug intervention, aortic aneurysm requiring surgical repair, any arterial thrombosis/embolism events, grade 3 or higher (Common Terminology Criteria for Adverse Events [CTCAE] 5.0) venous thrombosis/embolism events, transient cerebral ischemic attacks, cerebrovascular accidents;
* Abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation or intra-abdominal abscess within 6 months before the first study drug administration;
* Severe infection (CTCAE 5.0 > grade 2) occurred within 28 days before the first drug administration, such as severe pneumonia requiring hospitalization, bacteremia, infectious complications, etc.; active infection requiring intravenous anti-infection treatment within 2 weeks before the first drug administration or fever of unknown cause >38.5℃ (subject to the investigator's judgment, fever caused by the tumor can be enrolled);
* History of another primary malignant tumor, but malignant tumors that have been treated with curative treatment before the first intervention of the study and have no known active disease (more than 5 years) and a low potential for recurrence (such as skin basal cell carcinoma and skin squamous cell carcinoma treated with potential curative treatment) are excluded;
* History of gastrointestinal bleeding within 6 months before enrollment, or conditions judged by the investigator to have a risk of gastrointestinal bleeding (such as severe esophageal-gastric varices);
* Other severe physical or mental diseases or laboratory test abnormalities that may increase the risk of participating in the study, affect treatment compliance, or interfere with the study results, and patients judged by the investigator as unsuitable to participate in this study.

Exclusion Criteria:

* The subject requests to terminate study treatment;
* Disease progression occurs, and the investigator judges that continuing study treatment has no clinical benefit;
* Any clinical adverse event, laboratory test abnormality, or other medical condition occurs, making it likely that the subject will no longer benefit from continued medication；
* Pregnancy occurs in a female subject;
* There is a significant deviation from the protocol, and the investigator determines that study treatment should be terminated;
* The subject dies or is lost to follow-up;
* The study is terminated;
* Other situations determined by the investigator that require termination of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1115 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Defined as the time from the date of enrollment to the date of any recorded tumor progression or death from any cause.
Time to Progression (TTP) | 2 years
  Defined as the time from the date of enrollment to the date of any recorded tumor progression.
adverse events | 2 years
  Incidence and grading of adverse events (AE) and serious adverse events (SAE).

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Defined as the time from the start of patient enrollment to death from any cause.
Objective Response Rate (ORR) | 2 years
  Defined as the percentage of subjects with the best response of CR or PR among all subjects in the analysis dataset, from the first dose to the first record of disease progression or death from any cause (whichever occurs first), using the response evaluation criteria in solid tumors (RECIST 1.1 and mRECIST standards).
Disease Control Rate (DCR) | 2 years
  Defined as the percentage of subjects with the best response of CR, PR, or SD among all subjects in the analysis dataset, from the first dose to the first record of disease progression or death from any cause (whichever occurs first), using the response evaluation criteria in solid tumors (RECIST 1.1 and mRECIST standards).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai

IPD SHARING:
Plan to Share IPD: No